CLINICAL TRIAL: NCT06806033
Title: A Phase II, Open-Label, Multicenter Study to Evaluate the Optimization of the Cytokine Release Syndrome Profile for Glofitamab in Combination With Gemcitabine Plus Oxaliplatin in Patients With Relapsed/Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Study to Evaluate the Optimization of the Cytokine Release Syndrome Profile for Glofitamab in Combination With Gemcitabine Plus Oxaliplatin in Participants With Relapsed/Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO45434
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: B-Cell Non-Hodgkins Lymphoma
MeSH Terms: interventions — obinutuzumab; glofitamab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- R/R Aggressive B-Cell Non-Hodgkin's Lymphoma (Experimental): Participants with R/R aggressive B-cell Non-Hodgkin's Lymphoma will receive obinutuzumab pre-treatment, followed by glofitamab + gemcitabine + oxaliplatin, followed by glofitamab monotherapy.
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive intravenous (IV) obinutuzumab 7 days prior to the first dose of glofitamab.
Drug: Glofitamab — Participants will receive IV glofitamab, both in combination with gemcitabine and oxaliplatin and as monotherapy, for up to 12 cycles (cycle length = 21 days).
Drug: Gemcitabine — Participants will receive IV gemcitabine in combination with glofitamab and oxaliplatin for up to 8 cycles (cycles length = 21 days).
Drug: Oxaliplatin — Participants will receive IV oxaliplatin in combination with glofitamab and gemcitabine for up to 8 cycles (cycle length = 21 days).

SUMMARY:
The main goal of this trial is to study the frequency and severity of cytokine release syndrome (CRS) in participants with relapsed or refractory (R/R) aggressive B-cell Non-Hodgkin's lymphoma (DLBCL) who are using a combination of glofitamab + gemcitabine + oxaliplatin (Glofit-GemOx) followed by glofitamab-only treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed large B-cell lymphoma (de novo or transformed from FL) with one of the following diagnoses according to World Health Organization, fifth edition: DLBCL Not Otherwise Specified (NOS); High-Grade B-Cell Lymphoma (HGBL), NOS; DLBCL/HGBL with MYC and BCL2 rearrangements
* R/R disease, defined as: relapsed = disease that has recurred following a response that lasted >/= 6 months after completion of the last line of therapy; refractory = disease that did not respond to or that progressed < 6 months after completion of the last line of therapy
* At least one line of prior systemic therapy
* Participants who have failed only one prior line of therapy must not be a candidate for high-dose chemotherapy followed by autologous stem cell transplant (ASCT)
* At least one bi-dimensionally measurable (> 1.5 cm) nodal lesion, or one bi-dimensionally measurable (> 1 cm) extranodal lesion, as measured on CT scan
* Eastern Cooperative Oncology Group (ECOG) status of 0, 1, or 2
* According to the investigator's judgment, participants should be able to receive the step-up dose regimen in an outpatient setting
* Adequate hematologic and renal function

Exclusion Criteria:

* Prior enrollment in Studies GO41943 (NCT04313608), GO41944 (STARGLO; NCT04408638), or Study GO44900 (NCT06624085)
* Participant has failed only one prior line of therapy and is a candidate for stem cell transplantation
* Any history of Waldenstrom's macroglobulinemia
* Primary mediastinal B-cell lymphoma
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to obinutuzumab, gemcitabine or oxaliplatin, or tocilizumab
* Prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3
* Prior treatment with gemcitabine or oxaliplatin
* Peripheral neuropathy or paresthesia assessed to be Grade >/= 2 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 at enrollment
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to first study treatment
* Treatment with monoclonal antibodies for the purposes of treating cancer within 4 weeks prior to first study treatment
* Primary or secondary CNS lymphoma at the time of recruitment
* Prior CNS involvement that has been definitively treated and confirmed via magnetic resonance imaging (MRI) or cerebrospinal fluid analysis to be in complete remission is permissible
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* History of other primary malignancy, with exceptions defined by the protocol
* Significant or extensive cardiovascular disease
* Significant pulmonary disease (including moderate or severe obstructive pulmonary disease)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 4 weeks prior to the first study treatment
* Positive for: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); tuberculosis; hepatitis B virus (HBV); hepatitis C virus (HCV); chronic active Epstein-Barr viral infection
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH) or progressive multifocal leukoencephalopathy
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1 or better (with the exception of alopecia and anorexia)
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Prior solid organ transplantation or prior allogenic stem cell transplant
* Active autoimmune disease requiring treatment
* Prior treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor agents), within 4 weeks prior to first dose of study treatment
* Ongoing systemic corticosteroid use which, in the opinion of the investigator, puts the participant at increased risk of steroid-related iatrogenic adrenal insufficiency
* Recent major surgery (within 4 weeks before the first study treatment) other than for diagnosis
* Clinically significant history of cirrhotic liver disease
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the participant at high-risk from treatment complications
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 18 months after the final dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cytokine release syndrome (CRS) | Up to approximately 5 years

SECONDARY OUTCOMES:
Incidence of serious cytokine release syndrome (CRS) events | Up to approximately 5 years
CRS frequency relative to the start of glofitamab infusions | Up to approximately 5 years
Complete response (CR) rate as determined by independent review facility (IRF) and the investigator | Up to approximately 5 years
  CR rate is defined as the proportion of participants whose best overall response is a CR based on PET/CT according to the 2014 Lugano Response Criteria during the study, as determined by the Independent Review Facility and the investigator.
Overall response rate (ORR) as determined by IRF and the investigator | Up to approximately 5 years
  ORR is defined as the proportion of participants whose best overall response is a PR or a CR according to the 2014 Lugano Response Criteria during the study, as determined by the Independent Review Facility and the investigator.
Duration of response (DOR) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (Up to approximately 5 years)
  DOR is defined as the time from the first occurrence of a documented objective response (CR or PR) to disease progression, or death from any cause, whichever occurs first.
Duration of complete response (DOCR) | From the first occurrence of a documented CR to disease progression or death from any cause, whichever occurs first (Up to approximately 5 years)
  DOCR is defined as the time from the first occurrence of a documented CR to disease progression, or death from any cause, whichever occurs first.
Progression-free survival (PFS) as determined by the IRF and the investigator | From enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first (Up to approximately 5 years)
  PFS is defined as the time from enrollment to the first occurrence of disease progression according to the 2014 Lugano Response Criteria or death from any cause, whichever occurs first, as determined by the Independent Review Facility and investigator.
Overall survival (OS) | From enrollment to date of death from any cause (Up to approximately 5 years)
  OS is defined as the time from enrollment to date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hoffmann-La Roche
Locations (50):
- United States (30):
  - Alaska Oncology & Hematology, LLC, Anchorage, Alaska
  - Providence Medical Foundation, Fullerton, California
  - Los Angeles Cancer Network, Glendale, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - The Lundquist Institute for BioMedical Innovation at Harbor-UCLA Medical Cente, Torrance, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - North Florida/ South Georgia VA Medical Center, Gainesville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - St Luke?s Cancer Institute, Boise, Idaho
  - Cancer Care Specialists of Central Illinois, Swansea, Illinois
  - Mission Blood and Cancer - MercyOne Cancer Center, Waukee, Iowa
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Ctr, Baton Rouge, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - New York Oncology Hematology, P.C., Albany, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Oncology Associates of Oregon, P.C, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor Scott & White Health, Temple, Texas
  - Texas Oncology - Gulf Coast, The Woodlands, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates - Virginia Beach, Virginia Beach, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
- Epworth Hospital, East Melbourne, Victoria, Australia
- Canada (2):
  - Arthur J.E. Child Comprehensive Cancer Center, Calgary, Alberta
  - CancerCare Manitoba (CCMB), Winnipeg, Manitoba
- France (5):
  - CHU de Grenoble, La Tronche
  - Chu de Montpellier-St Eloi, Montpellier
  - CHU de Bordeaux, Pessac
  - CHU DE RENNES - CHU Pontchaillou, Rennes
  - Chu De Tours, Tours
- Germany (4):
  - CAMPUS BENJAMIN FRANKLIN CharitéCentrum 14 Med.Klinik f.Hämatologie u.Onkologie, Berlin
  - Charite-Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK), Berlin
  - Universitätsklinikum Köln, Cologne
  - Otto von Guericke Uni Magdeburg Uniklinik, Magdeburg
- Italy (5):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale, Napoli, Campania
  - IRCCS Istituto Romagnolo per lo studio dei tumori "Dino Amadori", Meldola, Emilia-Romagna
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili, Brescia, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing